CLINICAL TRIAL: NCT01534702
Title: Phase I/II Study on Cytarabine and Idarubicin Combined With Escalating Doses of Clofarabine as Induction Therapy in Patients With Acute Myeloid Leukemia and High Risk for Induction Failure (AMLSG 17-10)
Brief Title: Dose Escalation of Clofarabine in Combination With Cytarabine and Idarubicin as Induction Therapy in High Risk AML
Acronym: CIARA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Krauter, Professor of Medicine, Hannover Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KS-2009-003; 2010-021719-18 (EudraCT Number)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; chemotherapy; clofarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: clofarabine, cytarabine, idarubicin

INTERVENTIONS:
Drug: clofarabine, cytarabine, idarubicin — Treatment is stratified according to patients age (< 60 years vs. ≥ 60 years).
  Medication:
  Patients < 60 years:
  * idarubicin 7.5 mg/m2 iv, days 1 + 3
  * cytarabine 750 mg/m2 iv, days 1 to 5
  Patients ≥ 60 years:
  * idarubicine 6 mg/m2 iv, days 1 + 3
  * cytarabine 750 mg/m2 iv, days 1 to 5
  Clofarabine will be given in escalating doses to cohorts of at least three patients:
  Clofarabine:
  * level -1: 15 mg/m2 iv, days 1 to 5
  * level 1: 20 mg/m2 iv, days 1 to 5
  * level 2: 25 mg/m2 iv, days 1 to 5
  * level 3: 30 mg/m2 iv, days 1 to 5
  * level 4: 35 mg/m2 iv, days 1 to 5
  Patients will be recruited according to a 3+3 design. New cohorts will be initiated depending on toxicity of the previous cohort during the first induction cycle. Enrollment will begin with dose level 1.

SUMMARY:
With current chemotherapy protocols, in 60-80% of patients with acute myeloid leukemia (AML) the leukemic blasts in the bone marrow can be reduced to < 5%. This is called "complete remission (CR)" and is the prerequisite for cure of the disease. During the last years, several genetic and biologic risk factors for the achievement of CR have been defined, and the remission rates vary considerably between patient groups with different risk profiles. On one hand, patients with certain chromosomal or molecular aberrations have very high CR rates of approximately 90%. Moreover, in some of these patients, molecularly targeted therapies for specific genetic aberrations are currently evaluated in clinical trials. However, these genetic aberrations account for only 50-60% of the overall patient population in AML. The remaining patients have a significantly inferior CR rate of only 50-60% with 30% resistant disease after two cycles of standard induction chemotherapy. In conclusion, there is need for improved induction regimens in a large number of adult patients with AML. An improved CR rate in this patient population will increase the number of patients eligible for intensive consolidation such as an allogeneic stem cell transplantation and might thereby be the basis for a better overall outcome. However, there is no clear evidence that this goal can be achieved with the currently available chemotherapy protocols. Clofarabine (2-chloro-2-fluoro-deoxy-9-D-arabinofuranosyladenine) is a nucleoside analogon which combines properties of fludarabine and cladribine. Due to the lack of neurological side effects, clofarabine could be explored in higher doses than other nucleoside analogues and has shown considerable antileukemic activity in patients with relapsed or refractory acute leukemias and elderly AML patients alone or in combination with cytarabine. In addition, the combination of clofarabine, cytarabine and idarubicin has produced promising results with acceptable toxicity in patients with relapsed or refractory AML. Based on these initial studies, there is need for a further optimization of the clofarabine dose in this combination. The aim of the AMLSG 17-10 study is therefore to evaluate the tolerability and safety of increasing doses of clofarabine in combination with idarubicin/cytarabine in patients with high risk AML defined by the genetic and molecular risk profile.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed AML according to WHO classification and aged ≥ 18 years eligible for an intensive induction chemotherapy with with the following characteristics:

   * absence of a t(15;17), t(8;21), inv(16)/t(16;16) and the respective fusion transcripts PML-RARA, RUNX1-RUNX1T1 and CBFB-MYH11
   * absence of an activating FLT3-mutation (FLT3-ITD or TKD-mutation)
   * absence of an NPM1 exon12 mutation
2. Written informed consent
3. No previous cytotoxic chemotherapy for the treatment of AML (exception: oral hydroxyurea for up to 5 days during screening/baseline to control hyperleukocytosis)
4. Adequate renal and hepatic functions as indicated by the following laboratory values:

   * Serum creatinine > upper limit of normal (ULN) or glomerular filtration rate (GFR) > 60 mL/min/1.73 m2, respectively
   * Serum bilirubin < 1.5 x ULN
   * Aspartate aminotransferase (AST/SGOT)/ alanine aminotransferase (ALT/SGPT) < 2.5 x ULN
   * Alkaline phosphatase (ALP) < 2.5 x ULN
5. Capable of understanding the investigational nature, potential risks and benefits of the study
6. Women of childbearing potential must have a negative serum pregnancy test with a sensitivity of at least 25 MIU/ml within 72 hours prior to start of IMP treatment
7. Female patients must meet one of the following criteria:

   * For female patients > 50 years of age at the day of inclusion: Menopause since at least 1 year
   * Female patients < 50 years of age at the day of inclusion who meet all of the following criteria:

     * menopause since at least 1 year
     * serum FSH levels > 40 MIU/mL
     * serum estrogen levels < 30 pg/ml or negative estrogen test
   * 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral ovariectomy with or without hysterectomy
   * Correct use of two reliable contraception methods from the time of screening/baseline and during the study for a minimum of 90 days after the last administration of study medication. This includes every combination of a hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring) or of an intrauterine device (IUD) with a barrier method (diaphragm, cervical cap, Lea contraceptive, femidom or condom) or with a spermicide. In case the patient takes hormone preparations for suppression of menstruation during the period of aplasia, a suitable and effective method of contraception has to be discussed with the investigator and used by the patient
   * General sexual abstinence from the time of screening/baseline, during the study until a minimum of 90 days after the last administration of study medication
   * Having only female sexual partners
   * Monogamous relationship with sterile male partner
8. Male patients must meet one of the following criteria:

   * 6 weeks after surgical sterilization by vasectomy
   * Correct use of two reliable contraception methods from the time of screening/baseline and during the study for a minimum of 90 days after the last administration of study medication. This includes every combination of a hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring) or of an IUD with a barrier method (diaphragm, cervical cap, Lea contraceptive, femidom or condom) or with a spermicide.
   * General sexual abstinence from the time of screening/baseline, during the study until a minimum of 90 days after the last administration of study medication
   * Having only male sexual partners
   * Monogamous relationship with sterile female partner

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy or immunotherapy not defined in the study protocol
2. Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of oral hydroxyurea. The patient must have recovered from all non-hematological acute toxicities from any previous therapy
3. Participation in a clinical trial within 30 days before inclusion in this study or concurrent to this study.
4. Bleeding disorder independent of AML
5. Patients with uncontrolled systemic fungal, bacterial, viral or other infection (defined as persistent disease signs/symptoms without improvement despite appropriate antibiotics or other treatment)
6. HIV Infection
7. Pregnant or lactating women
8. Any significant concurrent disease, illness, psychiatric disorder or history of serious organ dysfunction that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
9. Diagnosis of another malignancy, unless the patient is disease-free for at least 3 years following the completion of curative intent therapy, with the following exceptions:

   * Myelodysplastic syndrome (MDS) in patients with AML after MDS according to the WHO classification
   * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
10. Known hypersensitivity to any of the investigational medical products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-04 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
maximal tolerated dose of clofarabine in combination with cytarabine and idarubicin | six weeks
  maximal tolerated dose of clofarabine in combination with cytarabine and idarubicin in the therapy of previously untreated AML and high risk for induction failure

SECONDARY OUTCOMES:
complete remission rate | 12 weeks
  complete remission rate after two cycles of induction therapy
relapse-free, event-free and overall survival | 4 years
blast reduction in the bone marrow after the first induction cycle | 15 days
duration of aplasia | 12 weeks
therapy-associated morbidity and mortality | 12 weeks
course of molecular and cytogenetic markers during chemotherapy | four years
  molecular and cytogenetic markers will be evaluated by cytognetic analysis and molecular techniuques (e.g. RT-PCR)
fraction of patients who receive an allogeneic stem cell transplantation in first complete remission | four years

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Krauter, MD, Principal Investigator — Hannover Medical School
Locations (7):
- Germany (7):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum Essen-Werden, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - Klinikum Rechts der Isar, München
  - Universitätsklinikum Ulm, Ulm